CLINICAL TRIAL: NCT02952196
Title: Cannabinoids as a New Intervention for Amphetamine Dependence: A Proof-of-concept Study
Brief Title: Cannabioids as a New Intervention for Amphetamine Dependence
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 16.181
Record Dates: First submitted 2016-10-27; First posted 2016-11-02 (Estimated); Last update posted 2020-10-23 (Actual); Status verified 2019-01

CONDITIONS: Amphetamine Addiction
Keywords: Amphetamine; Cannabinoids
MeSH Terms: conditions — Amphetamine-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- placebo (Placebo Comparator)
  Interventions: Drug: drug administration
- cannabinoid dose 1 (Experimental)
  Interventions: Drug: drug administration
- cannabinoid dose 2 (Experimental)
  Interventions: Drug: drug administration

INTERVENTIONS:
Drug: drug administration — administering drug to patient with amphetamine addiction

SUMMARY:
Addiction to amphetamine is characterized by alternating phases of intoxication and short abstinence, followed by recurrent drug-craving episodes which result in distress and relapse. Addiction involves a number of neurotransmission systems, including the endocannabinoid system (ECBS). It has been demonstarted that cannabidioids can have physiological, anxiolytic and neuroprotective properties. It has been shown to have multiple therapeutic properties for treating anxiety, schizophrenia and interestingly cannabinoids have been shown to be potentially helpful in treating addiction, due to their effects on various neuronal circuits involved in this disorder.

The investigators overall hypothesis is that cannabinoids are an interesting pharmacological contender to decrease amphetamine craving and treat amphetamine addiction.

ELIGIBILITY:
Inclusion Criteria:

* Current DSM-V criteria for amphetamine use disorder
* Ability to give valid, informed consent

Exclusion Criteria:

* Severe and/or unstable hepatic, neurologic (including diagnosis of seizures), cardiac (including arrhythmias) or renal disease, or any other severe or unstable medical condition that precludes safe participation in the study according to the study physician.
* Severe psychiatric condition (history of schizophrenia, schizoaffective disorder or bipolar disorder; current acute psychosis, mania or severe suicidality
* Any serious medical condition or psychiatric illness that precludes the subject from signing the informed consent form

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
assessing amphetamine craving | everyday during the study (that will last 3 days for each participants)
  using questionnaire to assess craving and taking vital signs

CONTACTS AND LOCATIONS:
Overall Officials: Didier Jutras-Aswad, MD, MS, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No